CLINICAL TRIAL: NCT00746980
Title: Efalizumab in the Treatment of Alopecia Totalis/Universalis in Young Adults, Phase II
Brief Title: Efalizumab in the Treatment of Alopecia, Phase II
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Newly identified safety concerns have changed the risk and benefit considerations
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology and Pediatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070823
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Alopecia Totalis
Keywords: alopecia; areata; universalis; severe; ophiasis; variants
MeSH Terms: conditions — Alopecia; Lymphoma, Follicular | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Subjects receiving drug
  Interventions: Drug: efalizumab

INTERVENTIONS:
Drug: efalizumab — 1 mg/kg subcutaneously once weekly for 48 weeks, following an initial conditioning dose of 0.7 mg/kg at week 0.
  Other Names: Raptiva

SUMMARY:
Determine the effect that treatment with efalizumab has on scalp hair re-growth in younger adults affected by severe variants of alopecia areata, including alopecia totalis, alopecia universalis, and severe ophiasis variants.

DETAILED DESCRIPTION:
This is a Phase II trial (single-center, open-label, prospective study) where subjects with severe forms of alopecia areata, namely alopecia totalis, universalis, and severe ophiasis, will be treated with efalizumab (Raptiva), a humanized monoclonal anti-CD11a antibody that reversibly inhibits T cell activation and migration, weekly for 48 weeks. We will assess for effect on hair and body re-growth as well as record any serious adverse events such as serious infections, thrombocytopenia, development of malignancy, and severe arthralgias to monitor for safety outcome data. Subjects will have regular physical examinations and laboratory studies throughout the study, as well as telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent and comply with study assessments for the full duration of the study.
* clinical diagnosis of alopecia totalis, alopecia universalis, or severe ophiasis variant of alopecia areata.
* 18-40 years of age.
* if a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception (birth control) for the duration of the study are necessary.
* if a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.

Exclusion Criteria:

* known hypersensitivity to efalizumab (Raptiva) or any of its components.
* known liver disease, including active hepatitis
* history of autoimmune diseases causing alopecia other than alopecia areata.
* prior biologic therapy within 6 months prior to study initiation.
* history of any malignancy within last ten years, except treated non-melanoma skin cancers.
* any woman currently pregnant or lactating.
* intake of systemic immunosuppressive agents, including oral corticosteroids, within 3 months prior to study initiation.
* history of positive PPD and/or tuberculosis.
* history of HIV/AIDS
* prior enrollment in any efalizumab study
* any condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* participation in another simultaneous clinical trial involving investigational agents.
* positive HIV screening test obtained at screening visit.
* positive QuantiFERON-TB test obtained at screening visit.
* positive hepatitis screen obtained at screening visit.
* platelet count 150 x 10(9)/L at baseline visit.
* presence of any abnormal laboratory value obtained at screening visit assessed as clinically significant by principal investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Percentage re-growth of scalp hair loss | 1 year

SECONDARY OUTCOMES:
Self-assessment (SA) and Static physician global assessment (SPGA) | 1 year
Body hair re-growth at 48 weeks | 1 year
Quality of life questionnaire | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis West, PhD, Principal Investigator — Northwestern University, Department of Dermatology